CLINICAL TRIAL: NCT05097807
Title: The Short-term and Long-term Impact of Word-picture-based and Short Video-based Shallow Reading Behavior in Social Media
Brief Title: The Impact of Shallow Reading in Social Media
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Principal Investigator, Wen Wang, MD & PhD, Director of radiology, Tang-Du Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 202103129
Record Dates: First submitted 2021-09-26; First posted 2021-10-28 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Social Media; Mental Health Disorder; Brain Imaging
Keywords: Social Media; Shallow reading; multimodal MRI; Brain network
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: Four parallel group, each with a different intervention, of which two are shallow reading in social media (different type), the other two are common use of smartphone.
Who Masked: Care Provider, Investigator
Masking Description: Participants know their intervention because they are informed to use their smartphone as expected.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- The impact of word-picture-based shallow reading in social media (Experimental): Use Microblog on their smartphone, a word-picture-based social media service similar to twitter.
  Interventions: Behavioral: smartphone related behaviors
- The impact of short video-based shallow reading in social media (Experimental): Use Tiktok on their smartphone, a short video-based social media service.
  Interventions: Behavioral: smartphone related behaviors
- The impact of full-length sci-fi novel reading (Active Comparator): Read a full-length sci-fi novel (Three body) on their own smartphone.
  Interventions: Behavioral: smartphone related behaviors
- The impact of film/TV series (Active Comparator): Watch a film on their own smartphone.
  Interventions: Behavioral: smartphone related behaviors

INTERVENTIONS:
Behavioral: smartphone related behaviors — Participants are required to watch specific contents on their own smartphones.

SUMMARY:
Social media is pervasively used in our life. There is a research hypothesis that the information in social media is "shallow" and the long-term use of it will cause readers' addiction, insomnia, and inability to pay attention, thus reducing the efficiency of learning and working. However, there is no systematic study on the relationship between "shallow reading" in social media and attention, addiction, sleep quality, and other mental health. Therefore, the investigators intend to explore the effect of "shallow reading" in social media on mental health based on about 300 healthy subjects by conducting questionnaire, cognitive scale assessment, multi-mode MRI scanning and EEG monitoring. A cross-sectional study will be combined with a longitudinal study to explore the clinical characteristics its relationship to brain function.

DETAILED DESCRIPTION:
With the development of social media such as "twitter", "Facebook" and "Microblog", "shallow reading" has gradually become the main way for people to obtain external information and relax. "Shallow reading" is characterized by incomplete and intermittent reading patterns, and readers often "dip into it" without thinking. There is a research hypothesis that the information in social media is "shallow" and the long-term use of it will cause readers' addiction, insomnia, and inability to pay attention, thus reducing the efficiency of learning and working. Some researchers even concern that "shallow reading" is destroying human beings' suspicion spirit, thinking ability and rational thinking which are based on writing and print culture. However, there is no systematic study on the relationship between "shallow reading" and attention or other mental health, not to mention its fMRI and EEG characteristics. Therefore, the investigators intend to explore the effect of "shallow reading" in social media on mental health based on about 300 healthy subjects by conducting questionnaire, cognitive scale assessment, multi-mode MRI scanning and EEG monitoring. A cross-sectional study will be combined with a longitudinal study to better understand both the short-term and long-term effect of "shallow reading" habit to the mental health and imaging characteristics. The collected indexes will be analyzed to explore the clinical characteristics of people with the habit of "shallow reading", and its relationship to mental health, brain imaging characteristics will finally be clarified.

ELIGIBILITY:
Inclusion Criteria:

1. Health volunteers
2. Capable to use smartphone

Exclusion Criteria:

1. Participants with a BMI greater than 30 or less than 18.5
2. Any use of cigarettes or alcohol
3. Color blindness
4. Left-handedness
5. With mental or psychiatric disorders
6. With cognitive impairment
7. Has a history of brain trauma
8. Has a family history of psychiatric disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Dynamic change of sustained attention from baseline state to after 2 hours of social media use | Baseline state and after 2 hours
  Continuous performance test (CPT) will be used to assess the difference of sustained attention before and after social media use.
  minimum: 0 maximum values: 1 Higher scores mean a better outcome.
Dynamic change of selective attention from baseline state to after 2 hours of social media use | Baseline state and after 2 hours
  Stroop color word test (SCWT) will be used to assess the difference of selective attention before and after social media use.
  minimum: 0 maximum values: 1 Higher scores mean a better outcome.

SECONDARY OUTCOMES:
Cerebral blood flow changes from baseline state to after 2 hours of social media use | Baseline state and after 2 hours
  Artery spin labeling (ASL) in MRI will be used to assess the difference of cerebral blood flow before and after social media use.
Brain functional connectivity changes from baseline state to after 2 hours of social media use | Baseline state and after 2 hours
  Blood oxygen level dependent (BOLD) in MRI will be used to assess the difference of functional connectivity before and after social media use.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Hu, MD, Principal Investigator — Department of Radiology, Fourth Military Medical University; YuTing Li, MD, Principal Investigator — Department of Radiology, Fourth Military Medical University; JingTing Sun, MD, Principal Investigator — Department of Radiology, Fourth Military Medical University; YuXuan Shang, MD, Principal Investigator — Department of Radiology, Fourth Military Medical University

IPD SHARING:
Plan to Share IPD: Yes
All demographic data, mental state assessments, and imaging data will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: All data will be open for other researchers after 5 years from the completion of data recruitment.
Access Criteria: Personal communication